CLINICAL TRIAL: NCT01665001
Title: Optimization of the Treatment of Adults With Precursor Lymphoid Neoplasms With Adjustment of the Type and Intensity of the Therapy for Age, Status of Minimal Residual Disease, Genetic and Phenotypic Features
Brief Title: Personalized Therapy of Precursor Lymphoid Neoplasms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice (Other)
Collaborators: Polish Adult Leukemia Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALG ALL6
Record Dates: First submitted 2012-08-11; First posted 2012-08-15 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Precursor Lymphoid Neoplasms
Keywords: Acute lymphoblastic leukemia; Induction; Consolidation; Minimal residual disease; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multiagent induction-consolidation (Experimental): Induction, consolidation, HSCT, maintenance for adults with newly diagnosed precursor lymphoid neoplasms
  Interventions: Other: Treatment strategy: induction, consolidation, HSCT, maintenance

INTERVENTIONS:
Other: Treatment strategy: induction, consolidation, HSCT, maintenance — Patients <55 years Ph-neg.: induction (daunorubicin, prednisone, vincristin, PEG-asparaginase), 2nd induction (if non-remission or MRD>0.1%; FLAM, MiniFLAM or FLAM-CAMP dependent on age and phenotype), consolidation (methotrexate, etoposide, cytarabine, cyclophosphamide, PEG-asparaginase). If MRD <0.01%: autoHSCT + maintenance (mercaptopurine, methotrexate) or multiagent maintenance (additionally daunorubicin, vincristin, prednisone); remaining patients: alloHSCT. Prophylaxis of leptomeningeal involvement: liposomal cytarabine intrathecally.
  Patients >55 years, Ph-neg.: as above, reduced doses. AlloHSCT with reduced conditioning.
  Patients Ph-pos.: as above, reduced doses in combination with continues imatinib. All intended for alloHSCT.

SUMMARY:
The primary goal of this study by The Polish Adult Leukemia Group (PALG) is to verify if individual therapeutic approach taking into account biological and phenotypic differences as well as response at the level of minimal residual disease is associated with improved outcome of adults with precursor lymphoid neoplasms

DETAILED DESCRIPTION:
Between 1997-2010 the PALG run three prospective studies. In the most recent PLAG 5-2007 protocol attempts have been made to individualize treatment. In particular, stratification to high and standard risk group was based on both conventional clinical criteria and the level of MRD after induction and consolidation. Patients with unsatisfactory response were referred for allogeneic hematopoietic stem cell transplantation (alloHSCT). Interim analysis showed significant improvement compared to previous PALG 4-2002 protocol with regard to both overall survival and leukemia-free survival. The reasons of failure were relapses and non-relapse mortality (NRM) associated with alloHSCT.

In the current protocol we intend to further adjust the therapy for individual patients needs. We assume that this way we will be able to reduce the risk of relapse and NRM and improve the cure rate. All patients will receive multiagent induction and consolidation chemotherapy. The type and intensity of the therapy, as well as indications for allogeneic and autologous HSCT will depend on age, status of MRD, immunophenotype and the presence of BCR/ABL fusion gene.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of PLN according to WHO 2008 classification
* Age ≥18 years
* Biological status allowing administration of induction therapy
* Informed patient consent form signed

Exclusion Criteria:

* Pregnancy
* Psychiatric diseases
* History of other malignancies
* HIV infection
* Active hepatitis
* Hypersensitivity to drugs used in induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | three years

SECONDARY OUTCOMES:
Leukemia-free survival | three years

OTHER OUTCOMES:
Remission duration | three years

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Giebel, MD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland

REFERENCES:
- [Background] Holowiecki J, Krawczyk-Kulis M, Giebel S, Jagoda K, Stella-Holowiecka B, Piatkowska-Jakubas B, Paluszewska M, Seferynska I, Lewandowski K, Kielbinski M, Czyz A, Balana-Nowak A, Krol M, Skotnicki AB, Jedrzejczak WW, Warzocha K, Lange A, Hellmann A. Status of minimal residual disease after induction predicts outcome in both standard and high-risk Ph-negative adult acute lymphoblastic leukaemia. The Polish Adult Leukemia Group ALL 4-2002 MRD Study. Br J Haematol. 2008 Jun;142(2):227-37. doi: 10.1111/j.1365-2141.2008.07185.x. Epub 2008 May 19. PMID 18492099
- See also: The Polish Adult Leukemia Goup — http://palg.witaj.pl